CLINICAL TRIAL: NCT06446102
Title: Bifurcation Coronary Lesion 0-0-1
Status: Completed | Type: Observational
Sponsor: RCF@ICPS (Other)
Responsible Party: Principal Investigator, Francesca SANGUINETI, Principal Investigator, GCS Ramsay Santé pour l'Enseignement et la Recherche
Other Study IDs: 23.02718.000229
Record Dates: First submitted 2024-05-17; First posted 2024-06-06 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Coronary Bifurcation Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Research Involving Human Persons (RIHP 3) focusing on the treatment of type 0-0-1 bifurcation lesions in routine practice. Multicenter Study.

To retrieve and analyze the details of different angioplasty techniques used in this type of bifurcation lesion (Medina 0-0-1) in order to describe current practice and search for predictors of clinical events.

DETAILED DESCRIPTION:
The primary objective of the trial is to estimate the frequency of Major Adverse Cardiac Events (MACE), including cardiac death, myocardial infarction within the territory of the treated lesion, and revascularization of the target lesion in a representative population of patients treated by coronary angioplasty of type 0-0-1 bifurcation lesions.

The sample size will be determined by the number of angioplasties of type 0-0-1 bifurcation lesions performed at each center between 2016 and 2022.

Since the trial is observational in nature and there are no previously published studies, the sample size cannot be calculated based on the desired precision of the estimation.

Furthermore, the purpose of the study is also to assess the techniques used to treat this type of coronary bifurcation and to highlight any differences between different centers and with other types of coronary bifurcation lesions described in the literature.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 years and older,
* Who underwent angioplasty for a coronary bifurcation lesion of type 0-0-1 between 2016 and 2022.

Exclusion Criteria:

- Opposing the collection and processing of necessary data and refusing additional telephone follow-up

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: In this trial, approximately 300 patients will be recruited from the Hôpital Privé Jacques Cartier in Massy, Clinique Pasteur in Toulouse, and Maasstad Hospital in Rotterdam between 2016 and 2022.
Sampling Method: Probability Sample
Enrollment: 273 (Actual)
Dates: Start 2023-12-11 (Actual); Primary Completion 2023-12-29 (Actual); Study Completion 2023-12-29 (Actual)

PRIMARY OUTCOMES:
Major Adverse Cardiovascular Events | 3 years
  Composite of cardiovascular death rate, myocardial infarction rate and target vessel revascularization rate.

SECONDARY OUTCOMES:
Target lesion revascularization | 3 years
  Target lesion revascularization rate

CONTACTS AND LOCATIONS:
Overall Officials: Francesca SANGUINETI, MD, Principal Investigator — ICPS
Locations (3):
- France (2):
  - Institut Cardiovasculaire Paris Sud, Hôpital Privé Jacques Cartier, Massy
  - Clinique Pasteur, Toulouse
- Maasstad Ziekenhuis, Rotterdam, Netherlands

DOCUMENTS (1):
  • Study Protocol (2023-10-16): https://cdn.clinicaltrials.gov/large-docs/02/NCT06446102/Prot_000.pdf